CLINICAL TRIAL: NCT05711836
Title: Role of HLA Genes and Innate Immunity in the Phenotypic Variability of COVID-19 an Italian, Prospective, Multicenter Association Study
Brief Title: Role of HLA Genes and Innate Immunity in the Phenotypic Variability of COVID-19
Acronym: 3490
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: HLA GENES
Record Dates: First submitted 2023-02-01; First posted 2023-02-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients
  Interventions: Genetic: HLA-genotyping
- controls
  Interventions: Genetic: HLA-genotyping

INTERVENTIONS:
Genetic: HLA-genotyping — HLA genotyping in DNA samples from peripheral blood of patients and controls

SUMMARY:
Case-control, prospective retrospective association study of patients infected with SARS-CoV2 and cured by COVID19. Recruited patients were divided into two cohorts (cases: patients with respiratory failure that required hospitalization and ventilatory assistance. Controls: patients who had oligo-asymptomatic forms of COVID19). Patients' blood samples were collected on bibula paper, from which genomic DNA was extracted. Next-generation sequencing of HLA and innate immunity genes was performed on these samples. Genetic risk and protective variants were identified, based on the distribution of allele frequencies in the two cohorts. The aim of the study is to evaluate the role of genes of the HLA system and innate immunity in modulating the host response to SARS-CoV2 infection. The identification of these factors is essential from the perspective of public health (identifying individuals most in need of protection from infection as they are at higher risk of severe forms), basic research (characterization of molecular mechanisms of disease) and therapeutics (through knowledge of basic mechanisms, identify potential therapeutic targets and optimize the protective efficacy of vaccines).

ELIGIBILITY:
Inclusion Criteria:

* Oxygen saturation (SaO2) <94% on room air; <90% if known chronic hypoxic conditions or receiving chronic supplemental oxygen
* Respiratory rate >24 breaths/min

Exclusion Criteria:

* Patients who still test positive for the presence of SARS-CoV-2 genome at the recruitment.
* Patients who cannot understand the meaning of the study and/or do not sign the informed consent form.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects healed from severe forms of COVID19 and oligo/asymptomatic subjects as controls
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Severe COVID19 | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Francesco Danilo Tiziano, Roma, Rm, Italy